CLINICAL TRIAL: NCT03277079
Title: Low Dose Statins, Ezetimibe and Nutraceuticals in Coronary Artery Disease Patients Intolerant to High Intensity Statin Treatment (TArget ChOlesterol)
Brief Title: Low Dose Statins, Ezetimibe and Nutraceuticals
Acronym: TACO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123/D/2017
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; LDL cholesterol; therapeutic target
MeSH Terms: conditions — Coronary Artery Disease | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- statin + ezetimibe (Active Comparator): Low dose statin associated with ezetimibe
  Interventions: Drug: statin + ezetimibe; Drug: statin + ezetimibe + Nutraceuticals
- statin + ezetimibe + Nutraceuticals (Active Comparator): Low dose statin associated with ezetimibe and Nutraceuticals
  Interventions: Drug: statin + ezetimibe; Drug: statin + ezetimibe + Nutraceuticals

INTERVENTIONS:
Drug: statin + ezetimibe — Combination of two drugs
  Other Names: Anticholesterol drug
Drug: statin + ezetimibe + Nutraceuticals — Combination of two grus plus nutraceuticals
  Other Names: Anticholesterol drug

SUMMARY:
It remains unknown if the association between moderate to low intensity statin therapy and ezetimibe and nutraceuticals might have a therapeutic role in high-intensity statin intolerant patients

DETAILED DESCRIPTION:
The aim of this study will be to evaluate whether the association between statin and exetimibe vs statin + ezetimibe + nutraceuticals can lead to higher percentage of LDL target achievement

ELIGIBILITY:
Inclusion Criteria:

Patients with angiographically assessed diagnosis of coronary artery disease

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic target | Up to 3 months
  LDL cholesterol < 70 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gaudio, MD, Study Chair — Sapienza University
Locations (1):
- Sapienza University, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marazzi G, Campolongo G, Pelliccia F, Calabro Md P, Cacciotti L, Vitale C, Massaro R, Volterrani M, Rosano G. Usefulness of Low-Dose Statin Plus Ezetimibe and/or Nutraceuticals in Patients With Coronary Artery Disease Intolerant to High-Dose Statin Treatment. Am J Cardiol. 2019 Jan 15;123(2):233-238. doi: 10.1016/j.amjcard.2018.09.041. Epub 2018 Oct 19. PMID 30420184